CLINICAL TRIAL: NCT04198077
Title: Conservative vs Conventional Oxygen Administration in Critically Ill Patients: Effects on ICU Mortality. A Multicentre Randomized Open Label Clinical Trial
Brief Title: Conservative Versus Conventional Oxygen Administration in Critically Ill Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Massimo Girardis, Head of Anesthesiology and Intensive Care Unit, University Hospital of Modena, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICUconservativeO2; 2018-002525-35 (EudraCT Number)
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Critical Illness; Respiration, Artificial; Hyperoxia; Hyperoxemia
Keywords: Mechanical Ventilation; Critically ill patient; Oxygenation; ICU; Intensive Care Unit
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration; Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: The study is designed as multicentre, open label, two parallel groups, randomized superiority clinical trial. The included patients will be randomized in 1:1 ratio in conservative and conventional group. A block randomisation will be used with variable block sizes (block size 4-6-8), stratified by center. Central randomisation will be performed using a secure, web-based, randomisation interface. The allocation sequence will be generated by the study statistician using computer generated random numbers.
Who Masked: Participant
Masking Description: The study is conceived as single blinded: only the patients will be not aware of the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONSERVATIVE (Experimental): Participants in the conservative group will receive the lowest FiO2 to maintain SpO2 between 94 and 98 percentage, or when available a PaO2 between 70 mmHg and 100 mmHg. A SpO2 alarm limit of 99 percent will apply whenever supplemental oxygen is being administered. The FiO2 will be reduced or oxygen supplementation discontinued whenever the SpO2 or PaO2 exceeded 98 percent or 100 mm Hg. An oxygen supplementation will be given only if SpO2 falls below 94 percent. Pre-oxygenation with FiO2 1.0 will not be performed during in-hospital transports or in anticipation of diagnostic and therapeutic manoeuvres.
  Interventions: Drug: Oxygen
- CONVENTIONAL (Active Comparator): In the conventional group, participants will receive a FiO2 aiming to maintain a SpO2 equal or major than 98 percentage, accepting an upper limit of PaO2 of 150 mmHg and a lower limit of 70 mmHg. The use of a FiO2 of less than 0.3 whilst ventilated is discouraged. According to standard Intensive Care Unit practice, control patients will receive a FiO2 of 1.0 during endotracheal intubation manoeuvre, airway suction or in-hospital transfers.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Administered via invasive or non-invasive mechanical ventilation with fraction of inspired oxygen between 0.21 and 1.0

SUMMARY:
Oxygen supplementation in the inspired mixture is commonly used in critically ill patients and observational studies highlight that those patients remain hyperoxemic for substantial periods during Intensive Care Unit stay. However, exposure to inhaled oxygen-enriched mixtures is widely recognized as potentially harmful and cause of organ damage. Although, the specific level of arterial oxygen partial pressure (PaO2) considered harmful, or the dangerous duration of hyperoxia, is not determined yet as there are no clinical trials on humans that evaluate the appropriate percentage of oxygen considered safe to maintain an adequate tissue oxygen availability.

The study is designed as a multicentre, open-label, two parallel groups, randomized superiority clinical trial. The study will involve 10 European intensive care units and will recruit adult critically ill patients requiring mechanical ventilation with an expected length of stay of more than 72 hours admitted to the Intensive Care Unit. Within the conventional group, participants will receive an inspired oxygen fraction (FiO2) aiming to maintain an oxygen saturation by pulse oximetry (SpO2) equal or major than 98 percentage, accepting an upper limit of PaO2 of 150 mmHg and a lower limit of 60 mmHg. Patients in the conservative group will receive the lowest FiO2 to maintain SpO2 between 94 and 98 percentage, or when available a PaO2 between 60 mmHg and 100 mmHg. The primary objective of this study is to verify the hypothesis that strict maintenance of normoxia improves survival in a wide population of mechanically ventilated critically ill patients compared to the application of conventional more liberal strategies of oxygen administration. Survival will be measured at Intensive Care Unit discharge.

The confirmation of the efficacy of a conservative strategy for oxygen administration in reducing the mortality rate among critically ill patients will lead to a profound revision of the current clinical practice and a rationale revision of the current recommendations would be mandatory, maybe also in other clinical scenarios such as emergency departments.

DETAILED DESCRIPTION:
Objectives: The primary objective of this study is to verify the hypothesis that strict maintenance of normoxia improves survival in a wide population of mechanically ventilated critically ill patients compared to the application of conventional more liberal strategies of oxygen administration. Survival will be measured at Intensive Care Unit discharge. Secondary objectives are to verify the hypothesis that, in a wide population of mechanically ventilated critically ill patients, the strict maintenance of normoxia compared to the application of conventional more liberal strategies of oxygen administration reduces the 90-day mortality, onset of new organ failures (respiratory, cardiovascular, renal and hepatic after 48 hours from Intensive Care Unit admission) during Intensive Care Unit stay, occurrence of nosocomial infections during Intensive Care Unit stay (only microbiologically documented bloodstream, respiratory and surgical site infections will be considered), the length of mechanical ventilation, vasopressor use and Intensive Care Unit stay, the occurrence of Intensive Care Unit acquired weakness and cognitive dysfunction.

Intervention: On the Intensive Care Unit admission, or later when they fulfil eligibility criteria, participants will be randomly assigned to a group of liberal conventional oxygen administration (CONVENTIONAL) or a group of conservative experimental oxygen administration (CONSERVATIVE). Within the conventional group, participants will receive a FiO2 aiming to maintain a SpO2 equal or major than 98 percentage, accepting an upper limit of PaO2 of 150 mmHg and a lower limit of 60 mmHg. Patients in the conservative group will receive the lowest FiO2 to maintain SpO2 between 94 and 98 percentage, or when available a PaO2 between 60 mmHg and 100 mmHg. The changes in oxygen therapy will be according to a nurse order-set. The indications to non-invasive ventilation or tracheal intubation and invasive mechanical ventilation (and to the most appropriate mode of ventilatory support) will be guided by principles of the Good Clinical Practice and by the clinical judgement of the attending physician. No other pharmacological therapy or treatment will be influenced by the study protocol. There are no restrictions to concomitant treatments provided to patients in this study.

Sample size and recruitment: Assuming a two-sided alpha level inferior than 0.05 and a power of 80 percentage, we calculated that 460 patients are needed per arm to detect a relative risk reduction of 40 percentage (absolute risk reduction of 6 percentage) compared to a mortality of 15 percentage observed in conventional group patients in previous studies. The global sample size is established to 1,000 patients. This includes an additional 80 participants to allow for drop-outs and an expected temporal trend of reducing mortality at ICU discharge. Every month, recruitment status will be evaluated, and a newsletter will be disseminated, including any issue arisen. The study will end after 12 months of enrollment plus 90 days for follow up.

Allocation and blinding: A block randomisation will be used with variable block sizes, stratified by centre using a web-based, randomisation interface.

Data collection and management: The study data will be collected along the entire Intensive Care Unit stay in a dedicated Case Report Form, that will be provided by the steering committee with proper options to minimize data entry errors: the data sheet will incorporate unmodifiable fixed intervals of values (for continuous variables) and pre-defined coding system (for binary or categorical variables). Data entry will be performed and double-checked from a dedicated researcher in each centre; in order to limit collection errors, 10 percent of all records will be randomly re-checked from the Principal Investigator in each participating centre. Data will be collected in an electronic Case report Form and transmitted by a dedicated platform to the Research and Innovation Office of the University Hospital of Modena protected by password to prevent unintentional modifications or deletion. Database management and quality control for this study will be under the responsibility of the Clinical Trial Quality Team of the University Hospital of Modena. In addition, each satellite centre will monthly communicate and report via e-mail with the coordinating centre about the number of recruited patients, eventual missing data or missing visit or any kind of problem correlated to data collection. Data related to the study will be stored for eventual further analysis or study purpose for 5 years after the end of the study. All the data about the included patients will be extrapolated from the clinical documentation and recorded in a Case Report Form from an adequately formed researcher. Demographic information (gender, age), co-morbidities, reason of Intensive Care Unit admission, type of admission will be registered at the inclusion; severity of critical illness (quantified by the Simplified Acute Physiology Score II) will be calculated by the data from the first 24 hours of Intensive Care Unit stay. During the entire stay, Sequential Organ Failure Assessment score will be calculated and registered daily. Every partial score will be registered separately (Nervous System, Respiratory, Cardiovascular, Liver, Renal and Coagulative). Blood Gas Analysis results will also be reported: FiO2, PaO2, PaCO2, hydrogen ion concentration, lactates, bicarbonates, Base Excess. Other daily parameters: duration of ventilatory support in hours, need and dose of vasoactive drugs (doses reported in µg/Kg/min), need of renal replacement therapy subsequent to the first 24 hours of Intensive Care Unit stay. The occurrence of Intensive Care Unit-acquired respiratory, blood and surgical site infections and the implicated microorganisms will be registered. Data from routine laboratory test will be reported: haemoglobin, platelets count, white blood cells count, coagulative parameters, parameters for liver and renal function; Central venous oxygen saturation and arterial lactates will be reported when available. The patient will be followed-up until 90 days and for patients who have been discharged from the hospital during this follow-up, the information will be collected with a phone interview. The vital status may be ascertained through public registries, in case of failure of all other ways of contact.

Statistical analysis: The intention to treat population will be considered for the primary analysis. A descriptive statistical analysis will be performed to describe every relevant variable. Kolmogorov-Smirnov normality test will be performed in order to verify the distribution of the variables. Results will be expressed in mean ± standard deviation or median and interquartile range as appropriate. Baseline and outcome variables will be compared between the two groups using the Mann-Whitney U test or t-test as appropriate. Categorical variables will be compared using Fisher's Exact test. The effect of conservative oxygen therapy on Intensive Care Unit and long-term mortality will be explored in the intention to treat population by a Kaplan-Meier analysis and Log-Rank for the hazard ratio. The primary and secondary outcomes will be also evaluated in pre-defined subgroups: quartile distribution of Simplified Acute Physiology Score II and Sequential Organ Failure Assessment score (total and for single organ) at admission, patients with respiratory Sequential Organ Failure Assessment score equal or major than 3 (respiratory dysfunction), patients with cardiovascular Sequential Organ Failure Assessment score equal or major than 3 (shock), surgical admissions compared to non-surgical admissions, documented infections at admission and distribution of length of stay in Intensive Care Unit. The relationship between oxygen exposure and Intensive Care Unit mortality will be evaluated according to the quartile distribution of the median value of the daily Intensive Care Unit time-weighted PaO2 values. Every test will be performed considering a two-sided p-value inferior of 0,05 for statistical significance.

Data monitoring: An independent Data Safety Monitoring Board, consisting of 2 experts in clinical research in intensive care and 1 bio-statistic will be established before patient enrolment. The Data Safety Monitoring Board Charter will be prepared by the steering committee and signed by the members of the Data Safety Monitoring Board before the trial commences. The Data Safety Monitoring Board will receive a study report every 3 months starting from the first enrolled patient and will have access to all results and make the appropriate considerations about the appropriateness of the sample size, the efficiency and quality of data collection system. No stopping rules are foreseen, either for utility or for efficacy. Moreover, the Data Safety Monitoring has the right to stop the trial for safety reasons.

Safety: Throughout the course of the study, every effort must be made to remain alert to possible Adverse Events. If this occurs, the first concern should be for the safety of the subject. The Investigator's responsibilities include the following: (a) Daily monitoring of all Adverse Events and laboratory abnormalities, regardless of the severity or relationship to study treatment. Only Serious Adverse events will be reported to the Steering Committee and, then, to Data Safety Monitoring Board and Research and Innovation Office of the University Hospital of Modena; (b) Determine the seriousness, relationship, and severity of each Adverse Event; (c) Determine the onset and resolution dates of each event; (d) Report each serious event by fax or email to the Steering Committee and, then, to Data Safety Monitoring Board and Research and Innovation Office of the University Hospital of Modena within 24 hours of the study site staff becoming aware of the event; ( e) Pursue Serious Adverse Events follow-up information actively and persistently. Follow-up information must be reported to the Steering Committee within 24 hours of the study site staff becoming aware of new information and entered in the electronic Case Report Form; (f) Ensure all Serious Adverse Event reports in the electronic Case Report Form are supported by documentation in the subjects' medical records.

Ethics approval: The entire study protocol, including informative material for the patients and modules for the informed consent, will be evaluated from the Local Ethics Committee from the coordinating centre and from all the collaborating centres. Every intention to modify any element of the original protocol after the first approval will be promptly notified to the Ethics Committee and will be applicated only after its written authorization.

Consent and confidentiality: A written informed consent will be asked to each eligible patient before enrolment. If the patient will be unable to comprehend or to give his consent (because of compromised neurological status), the following consent options are acceptable: (a) A priori consent by a substitute decision-maker; (b) delayed consent from a substitute decision-maker; (c) Delayed consent from the patient; (d) waiver of consent; (e) consent provided by an ethics committee or other legal authority. Which options are available at individual participating sites will be determined by the relevant ethics committee and subject to applicable laws. Every patient is free to leave the study protocol at any stage of the study and can request to retire his consent and, consequently, to ask the elimination of all his data from the database. Data about personal and private information, included sensible data, will be treated following current legislation on data protection; patients will be identified with a coding system and data registered in an anonymous form.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients admitted to participant Intensive Care Units
* Age major than 18 years without regards about sex and ethnicity
* Expected length of Intensive Care Unit stay of more than 72 hours
* Need of any respiratory support (invasive or non invasive mechanical ventilation) at admission and with an expected length of respiratory support major than 6 hours
* Acquisition of informed consent

Exclusion Criteria:

* Pregnancy
* Admission to Intensive Care Unit after elective surgery
* Intensive Care Unit readmission (after a first discharge) in the study period
* Invasive or non invasive mechanical ventilation greater than 12 hours in the 28 days before study inclusion
* Clinical decision to withhold life-sustaining treatment or "too sick to benefit" or patients with a life expectancy of less than 28 days due to a chronic or underlying medical condition
* Previous enrolment in other interventional studies of targeted oxygen therapy
* Acute respiratory failure on chronic obstructive pulmonary disease
* Acute respiratory distress syndrome with a PaO2/FiO2 ratio less than 150
* Long-term supplemental oxygen therapy
* Patients candidate to hyperoxia treatment for reasons including (but not limited to) carbon monoxide poisoning or to hyperbaric oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-12-04 (Estimated); Study Completion 2023-03-04 (Estimated)

PRIMARY OUTCOMES:
Mortality | Intensive Care Unit discharge censored at day 90
  Intensive Care Unit mortality rate, defined as the number of deaths for any cause

SECONDARY OUTCOMES:
90-day mortality | At day 90 from admission
  Mortality for any cause
Occurrence of new organ dysfunction | From ≥48 hours after ICU admission to ICU discharge, censored at day 90
  Occurrence of new organ dysfunction during ICU stay. Organ dysfunction is defined as a Sequential Organ Failure Assessment (SOFA) score ≥3 for the corresponding organ occurring after randomization. SOFA score ranges from 0 (no organ dysfunction) to 24 (multiple organ failure)
Infections | From ≥48 hours after ICU admission to ICU discharge, censored at day 90
  Bloodstream, respiratory and surgical site infections defined according to the Centers for Disease Control and Prevention definition, only when microbiologically documented
Ventilation-free hours (VFHs) | From randomisation to ICU discharge, censored at day 90
  Total number of hours of unassisted breathing. Periods of assisted breathing lasting less than 24 hours for surgical procedures will not count against the calculation. Patients who are receiving extracorporeal membrane oxygenation will be defined as receiving assisted breathing irrespective of whether they are ventilated or not
Vasopressor free-hours | From randomisation to ICU discharge, censored at day 90
  Total number of hours without vasoactive drugs infusion used for hypotension
Intensive Care Unit free days at 28-day | From randomisation until day 28
  Days in which the patient is not in Intensive Care Unit
ICU free days at 90-day | From randomisation until day 90
  Days in which the patient is not in Intensive Care Unit
Cognitive Dysfunction | Measured at Intensive care Unit discharge (censored at day 90)
  Assessed by Mini-Mental State Examination Test ranging from zero (severe cognitive dysfunction ) to 30 (no cognitive dysfunction)
ICU acquired weakness | Measured at Intensive care Unit discharge(censored at day 90)
  ICU acquired weakness is defined by Medical Research Council (MRC) scale, when weakness had developed after ICU admission, is symmetric and the average MRC score is <4

CONTACTS AND LOCATIONS:
Locations (1):
- Girardis Massimo, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nash G, Blennerhassett JB, Pontoppidan H. Pulmonary lesions associated with oxygen therapy and artificial ventilation. N Engl J Med. 1967 Feb 16;276(7):368-74. doi: 10.1056/NEJM196702162760702. No abstract available. PMID 6017244
- [Background] Crapo JD, Hayatdavoudi G, Knapp MJ, Fracica PJ, Wolfe WG, Piantadosi CA. Progressive alveolar septal injury in primates exposed to 60% oxygen for 14 days. Am J Physiol. 1994 Dec;267(6 Pt 1):L797-806. doi: 10.1152/ajplung.1994.267.6.L797. PMID 7810684
- [Background] Pagano A, Barazzone-Argiroffo C. Alveolar cell death in hyperoxia-induced lung injury. Ann N Y Acad Sci. 2003 Dec;1010:405-16. doi: 10.1196/annals.1299.074. PMID 15033761
- [Background] Dieperink HI, Blackwell TS, Prince LS. Hyperoxia and apoptosis in developing mouse lung mesenchyme. Pediatr Res. 2006 Feb;59(2):185-90. doi: 10.1203/01.pdr.0000196371.85945.3a. PMID 16439576
- [Background] Bhandari V, Elias JA. Cytokines in tolerance to hyperoxia-induced injury in the developing and adult lung. Free Radic Biol Med. 2006 Jul 1;41(1):4-18. doi: 10.1016/j.freeradbiomed.2006.01.027. Epub 2006 Feb 17. PMID 16781448
- [Background] Baleeiro CE, Christensen PJ, Morris SB, Mendez MP, Wilcoxen SE, Paine R 3rd. GM-CSF and the impaired pulmonary innate immune response following hyperoxic stress. Am J Physiol Lung Cell Mol Physiol. 2006 Dec;291(6):L1246-55. doi: 10.1152/ajplung.00016.2006. Epub 2006 Aug 4. PMID 16891399
- [Background] Baleeiro CE, Wilcoxen SE, Morris SB, Standiford TJ, Paine R 3rd. Sublethal hyperoxia impairs pulmonary innate immunity. J Immunol. 2003 Jul 15;171(2):955-63. doi: 10.4049/jimmunol.171.2.955. PMID 12847267
- [Background] Orbegozo Cortes D, Puflea F, Donadello K, Taccone FS, Gottin L, Creteur J, Vincent JL, De Backer D. Normobaric hyperoxia alters the microcirculation in healthy volunteers. Microvasc Res. 2015 Mar;98:23-8. doi: 10.1016/j.mvr.2014.11.006. Epub 2014 Nov 26. PMID 25433297
- [Background] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Hogdall C, Lundvall L, Svendsen PE, Mollerup H, Lunn TH, Simonsen I, Martinsen KR, Pulawska T, Bundgaard L, Bugge L, Hansen EG, Riber C, Gocht-Jensen P, Walker LR, Bendtsen A, Johansson G, Skovgaard N, Helto K, Poukinski A, Korshin A, Walli A, Bulut M, Carlsson PS, Rodt SA, Lundbech LB, Rask H, Buch N, Perdawid SK, Reza J, Jensen KV, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Effect of high perioperative oxygen fraction on surgical site infection and pulmonary complications after abdominal surgery: the PROXI randomized clinical trial. JAMA. 2009 Oct 14;302(14):1543-50. doi: 10.1001/jama.2009.1452. PMID 19826023
- [Background] Stub D, Smith K, Bernard S, Bray JE, Stephenson M, Cameron P, Meredith I, Kaye DM; AVOID Study. A randomized controlled trial of oxygen therapy in acute myocardial infarction Air Verses Oxygen In myocarDial infarction study (AVOID Study). Am Heart J. 2012 Mar;163(3):339-345.e1. doi: 10.1016/j.ahj.2011.11.011. PMID 22424003
- [Background] Ballard C, Jones E, Gauge N, Aarsland D, Nilsen OB, Saxby BK, Lowery D, Corbett A, Wesnes K, Katsaiti E, Arden J, Amoako D, Prophet N, Purushothaman B, Green D. Optimised anaesthesia to reduce post operative cognitive decline (POCD) in older patients undergoing elective surgery, a randomised controlled trial. PLoS One. 2012;7(6):e37410. doi: 10.1371/journal.pone.0037410. Epub 2012 Jun 15. PMID 22719840
- [Background] Floyd TF, Clark JM, Gelfand R, Detre JA, Ratcliffe S, Guvakov D, Lambertsen CJ, Eckenhoff RG. Independent cerebral vasoconstrictive effects of hyperoxia and accompanying arterial hypocapnia at 1 ATA. J Appl Physiol (1985). 2003 Dec;95(6):2453-61. doi: 10.1152/japplphysiol.00303.2003. Epub 2003 Aug 22. PMID 12937024
- [Background] Tolias CM, Reinert M, Seiler R, Gilman C, Scharf A, Bullock MR. Normobaric hyperoxia--induced improvement in cerebral metabolism and reduction in intracranial pressure in patients with severe head injury: a prospective historical cohort-matched study. J Neurosurg. 2004 Sep;101(3):435-44. doi: 10.3171/jns.2004.101.3.0435. PMID 15352601
- [Background] Chiu EH, Liu CS, Tan TY, Chang KC. Venturi mask adjuvant oxygen therapy in severe acute ischemic stroke. Arch Neurol. 2006 May;63(5):741-4. doi: 10.1001/archneur.63.5.741. PMID 16682544
- [Background] Karu I, Loit R, Zilmer K, Kairane C, Paapstel A, Zilmer M, Starkopf J. Pre-treatment with hyperoxia before coronary artery bypass grafting - effects on myocardial injury and inflammatory response. Acta Anaesthesiol Scand. 2007 Nov;51(10):1305-13. doi: 10.1111/j.1399-6576.2007.01444.x. PMID 17944632
- [Background] Pryor KO, Fahey TJ 3rd, Lien CA, Goldstein PA. Surgical site infection and the routine use of perioperative hyperoxia in a general surgical population: a randomized controlled trial. JAMA. 2004 Jan 7;291(1):79-87. doi: 10.1001/jama.291.1.79. PMID 14709579
- [Background] Belda FJ, Aguilera L, Garcia de la Asuncion J, Alberti J, Vicente R, Ferrandiz L, Rodriguez R, Company R, Sessler DI, Aguilar G, Botello SG, Orti R; Spanish Reduccion de la Tasa de Infeccion Quirurgica Group. Supplemental perioperative oxygen and the risk of surgical wound infection: a randomized controlled trial. JAMA. 2005 Oct 26;294(16):2035-42. doi: 10.1001/jama.294.16.2035. PMID 16249417
- [Background] Suzuki S, Eastwood GM, Peck L, Glassford NJ, Bellomo R. Current oxygen management in mechanically ventilated patients: a prospective observational cohort study. J Crit Care. 2013 Oct;28(5):647-54. doi: 10.1016/j.jcrc.2013.03.010. Epub 2013 May 15. PMID 23683560
- [Background] Young PJ, Beasley RW, Capellier G, Eastwood GM, Webb SA; ANZICS Clinical Trials Group and the George Institute for Global Health. Oxygenation targets, monitoring in the critically ill: a point prevalence study of clinical practice in Australia and New Zealand. Crit Care Resusc. 2015 Sep;17(3):202-7. PMID 26282259
- [Background] Brower RG, Lanken PN, MacIntyre N, Matthay MA, Morris A, Ancukiewicz M, Schoenfeld D, Thompson BT; National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med. 2004 Jul 22;351(4):327-36. doi: 10.1056/NEJMoa032193. PMID 15269312
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] de Jonge E, Peelen L, Keijzers PJ, Joore H, de Lange D, van der Voort PH, Bosman RJ, de Waal RA, Wesselink R, de Keizer NF. Association between administered oxygen, arterial partial oxygen pressure and mortality in mechanically ventilated intensive care unit patients. Crit Care. 2008;12(6):R156. doi: 10.1186/cc7150. Epub 2008 Dec 10. PMID 19077208
- [Background] Girardis M, Busani S, Damiani E, Donati A, Rinaldi L, Marudi A, Morelli A, Antonelli M, Singer M. Effect of Conservative vs Conventional Oxygen Therapy on Mortality Among Patients in an Intensive Care Unit: The Oxygen-ICU Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1583-1589. doi: 10.1001/jama.2016.11993. PMID 27706466
- [Background] Setsukinai K, Urano Y, Kakinuma K, Majima HJ, Nagano T. Development of novel fluorescence probes that can reliably detect reactive oxygen species and distinguish specific species. J Biol Chem. 2003 Jan 31;278(5):3170-5. doi: 10.1074/jbc.M209264200. Epub 2002 Nov 4. PMID 12419811
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Kleyweg RP, van der Meche FG, Schmitz PI. Interobserver agreement in the assessment of muscle strength and functional abilities in Guillain-Barre syndrome. Muscle Nerve. 1991 Nov;14(11):1103-9. doi: 10.1002/mus.880141111. PMID 1745285
- [Background] Cook D, Lauzier F, Rocha MG, Sayles MJ, Finfer S. Serious adverse events in academic critical care research. CMAJ. 2008 Apr 22;178(9):1181-4. doi: 10.1503/cmaj.071366. No abstract available. PMID 18427095